CLINICAL TRIAL: NCT04720807
Title: Letrozole Combined With Anlotinib Hydrochloride in the Treatment of Platinum-resistant Recurrent Ovarian Cancer: a Prospective, Single-arm, Open Label, Exploratory Phase 2 Clinical Trial.
Brief Title: Letrozole Combined With Anlotinib Hydrochloride in the Treatment of Platinum-resistant Recurrent Ovarian Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XH-21-001
Record Dates: First submitted 2021-01-14; First posted 2021-01-22 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: Platinum-resistant Recurrent Ovarian Cancer

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Letrozole combined with anlotinib hydrochloride (Experimental): Letrozole combined with anlotinib hydrochloride in the treatment of platinum-resistant recurrent ovarian cancer.
  Interventions: Drug: Letrozole combined with anlotinib hydrochloride

INTERVENTIONS:
Drug: Letrozole combined with anlotinib hydrochloride — Letrozole combined with anlotinib hydrochloride in the treatment of platinum-resistant recurrent ovarian cancer.

SUMMARY:
The study is a prospective, single-arm, open label, exploratory phase 2 clinical trial, which aims to study the therapeutic effect of letrozole combined with anlotinib hydrochloride in platinum-resistant recurrent ovarian cancer.

DETAILED DESCRIPTION:
The study is a prospective, single-arm, open label, exploratory phase 2 clinical trial, which aims to study the therapeutic effect of letrozole combined with anlotinib hydrochloride in platinum-resistant recurrent ovarian cancer.The patient has undergone surgery and received ≥2 lines of platinum-containing chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older;
2. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2;
3. Histologically diagnosed epithelial ovarian cancer (high-grade serous, clear cell, endometrioid ovarian cancer), fallopian tube cancer or primary peritoneal cancer;
4. The patient has undergone surgery and received ≥2 lines of platinum-containing chemotherapy. During the treatment period of the platinum-containing regimen (from the beginning of the treatment to 1 month after the last chemotherapy), the curative effect is non-PD, and the disease relapse/progress within 6 months after the treatment；
5. The patient has measurable lesions with imaging evidence;
6. The expected survival period ≥ 3 months;
7. Estrogen receptor (ER) is positive in immunohistochemistry of the first or the last surgical specimens;
8. Adequate organ function at screening:

1) Adequate bone marrow function at screening: Hemoglobin ≥90 g/L (no blood transfusion within 14 days); Neutrophil ≥1.5×109/L; Platelets ≥80×109/L; 2) Biochemical test: Total bilirubin≤1.5×ULN (upper limit of normal); Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≤ 2.5×ULN; if there is liver metastasis, ALT or AST ≤ 5×ULN; Serum creatinine ≤ 1.5×ULN or endogenous creatinine clearance ≥ 50ml/min (Cockcroft-Gault formula); 9. The patient has not been treated with other tyrosine kinase inhibitor (TKI) drugs; 10. The patient has not received tumor endocrine therapy; 11. Patients should have good compliance and the family members agree to cooperate in the survival follow-up.

Exclusion Criteria:

1. Patients with other malignant tumors at the same time except for recovery or tumors in a stable state.
2. Pregnant or breast feeding women;
3. Patients participated in other drug clinical trials within six months;
4. Patients with many factors that affect oral drugs (such as inability to swallow, chronic diarrhea, intestinal obstruction, etc.);
5. Any bleeding event with a severity level of grade ≥ 3 in CTCAE 4.0 in the 4 weeks before screening;
6. Patients with known central nervous system metastasis or a history of the metastasis before screening;
7. Patients with hypertension who cannot be well controlled by antihypertensive drugs (systolic blood pressure> 140 mmHg, diastolic blood pressure> 90 mmHg); those with a history of unstable angina; those who are newly diagnosed with angina within 3 months before screening or Myocardial infarction occurred within 6 months before screening; arrhythmia requires long-term use of antiarrhythmic drugs and New York Heart Association grade ≥ II cardiac insufficiency;
8. Long-term unhealed wounds or incomplete fractures;
9. A previous history of organ transplantation;
10. Imaging shows that the tumor has invaded important blood vessels or the researcher has judged that the patient's tumor is highly likely to invade important blood vessels to induce fatal bleeding during treatment;
11. Abnormal coagulation function (PT>16s, APTT>43s, TT>21s, Fbg<2g/L); those with bleeding tendency (INR is normal without using anticoagulants in 14 days before randomization); patients treated with anticoagulants or vitamin K antagonists such as warfarin, heparin or their analogs; under the condition of INR ≤ 1.5, Low-dose warfarin (1 mg orally, once a day) or low-dose aspirin (do not exceed 100 mg per day) is permitted for preventive purposes;
12. Arteriovenous thrombosis events occurred within one year before screening, such as cerebrovascular accidents (including temporary ischemic attacks), deep vein thrombosis (venous thrombosis caused by intravenous catheterization due to pre-chemotherapy, except those who have been cured), and pulmonary embolism;
13. Those who have a history of psychotropic drug abuse and can't be prevented or have mental disorders;
14. Have a history of immunodeficiency, or have a history of organ transplantation;
15. According to the judgment of the investigator, there are accompanying diseases that seriously endanger the safety of the patient or affect the completion of the study;
16. Have a history of surgery within 28 days;
17. A history of abdominal fistula or gastrointestinal perforation within 28 days;
18. People who may receive other systemic anti-tumor treatments or plan to undergo ovarian cancer reduction surgery during the study period.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2022-08-31 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
ORR | 3 years
  objective response rate

SECONDARY OUTCOMES:
PFS | 3 years and 5 years
  progression-free survival time
OS | 3 years and 5 years
  Overall survival
AE | 3 years and 5 years
  Adverse event

CONTACTS AND LOCATIONS:
Locations (1):
- Xinhua Hospital Affiliated to Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality, China